CLINICAL TRIAL: NCT04781725
Title: A Phase II Randomized Window of Opportunity Trial Evaluating Clinical and Biological Effects of Intratumoral INT230-6 in Early Stage Breast Cancer: The INVINCIBLE Trial
Brief Title: INVINCIBLE TRIAL: Intratumoral INT230-6 in Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Intensity Therapeutics, Inc. (Industry); Ontario Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OTT 20-11 (IT-02)
Record Dates: First submitted 2021-01-25; First posted 2021-03-04 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: window of opportunity; intratumoral; Ki67; complete pathologic response (PCR); immune activation; INT230-6; cisplatin; vinblastine; cell cycle arrest
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response | interventions — Cisplatin; Vinblastine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- INT230-6 Treated Arm (Experimental): Part I: Patients will receive up to 3 doses of INT230-6 injected weekly prior to breast surgery
  Part II: Patients will receive up to 2 intratumoral doses of INT230-6 (over a 15-day period) prior to breast surgery
  Interventions: Drug: INT230-6; Other: Saline injection
- Control Arm (Placebo Comparator): Part I: No intervention while awaiting surgery
  Part II: Placebo saline injection
  Interventions: Other: Saline injection

INTERVENTIONS:
Drug: INT230-6 — INT230-6 is a formulation of two well known chemotherapeutic agents, cisplatin (0.5mg/mL) and vinblastine sulfate (0.1mg/mL), combined with 2-hydroxybenzoylaminooctanoate (also known as SHAO-FA or SHAO as a sodium salt at 10mg/mL).
  Other Names: Cisplatin; Vinblastine; 2-hydroxybenzoylaminooctanoate (SAHO)
  Arms: INT230-6 Treated Arm
Other: Saline injection — Standard 0.9 % NaCl Normal Saline

SUMMARY:
This is a phase II, randomized, multi-center, parallel design, window of opportunity trial evaluating intratumoral INT230-6 in up to 90 patients with early stage breast cancer. In a 2:1 randomization, patients on the treatment arm will receive intratumoral INT230-6 injections prior to breast surgery.

DETAILED DESCRIPTION:
The study comprises 2 consecutive parts. The first part will be to test safety and feasibility of the dosing procedures. Results from Part I of the study will standardise the optimal dose and frequency of INT230-6 for participants in Part II.

Part I: Open-label 2:1 randomized study of up to 30 patients. Treatment arm patients will be given up to 3 doses of INT230-6 injected weekly prior to breast surgery, at a dose based on longest diameter. The control arm patients receive no treatment.

Part II: Double-blind, 2:1 randomized study of up to an additional 60 patients. The placebo arm includes a saline injection of similar dose and frequency as the treatment arm (up to 2 doses of INT230-6/saline injected weekly prior to breast surgery).

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with newly diagnosed histologically confirmed primary invasive breast cancer currently not undergoing any treatment while awaiting surgery.
2. Patients with early, operable stage I to II breast cancer amendable for complete surgical resection as assessed by treating surgical oncologist.
3. Tumors must be clinically palpable by surgeon. Part I: ≥ 1.0 cm by palpation or on imaging. Part II: ≥ 1.5 cm by palpation or on imaging.
4. Histologic Bloom Richardson grade ≥2.

4. Invasive ductal or lobular carcinoma, invasive carcinoma Not Otherwise Specified (NOS).

5. ECOG PS 0-2 (Appendix A). 6. The participant (or legally acceptable representative if applicable) is able to provide written informed consent for the study.

Exclusion Criteria:

1. Locally advanced or metastatic breast cancer.
2. Prior therapy with chemotherapy or planned neoadjuvant chemotherapy.
3. Pre-dominant histology other than invasive ductal or lobular carcinoma or invasive carcinoma NOS.
4. Patients with an active infection.
5. Absolute Neutrophil Count < 1.5 x 10^9/L.
6. Patients with pre-existing renal impairment, Creatinine clearance calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation of less than 50 mL/min/1.73m2.
7. Any serious known immediate or delayed hypersensitivity reaction(s) to vinblastine or cisplatin or idiosyncrasy to drugs chemically related to the investigational drugs.
8. Known allergic reaction to local anesthetic (Xylocaine, Marcaine).
9. Concurrent medical condition requiring the use of immunosuppressive medications, or systemic corticosteroids at doses of greater than 10 mg Prednisone-equivalent Topical steroids and other localized corticosteroids are permitted. Use of steroids as prophylactic treatment for subjects with contrast allergies to diagnostic imaging contrast dyes will be permitted.
10. Concurrent use of a prohibited medication or planned use of any forbidden medications during treatment with INT230-6, or within 4 weeks prior to study drug administration, which include chemotherapy, immunotherapy (tumor vaccine, cytokine, or growth factor given to control the cancer: systemic or intratumoral), other biologic therapy, investigational therapy, or hormonal therapy, cisplatin containing agents, and vinblastine containing agents while on treatment in this study. Other prohibited concomitant medications that will interact with vinblastine and cisplatin include mitomycin, phenytoin, CYP3A4 inhibitors (ketoconazole, voriconazole, clarithromycin, erythromycin), nephrotoxic drugs (aminoglycosides, amphotericin), or pure pyridoxine (pyridoxine contained in multivitamin is permitted). Use of other investigational drugs (drugs not marketed for any indication) within 4 weeks prior to study drug administration not permitted.
11. Pregnancy if patient is of childbearing age) or breast feeding.
12. Subjects with signs/symptoms suggestive of COVID-19 or known COVID-19 positive contacts in the past 14 days would be tested as per local Public Health and/or Institutional Guidelines. If patients are COVID-19 positive at the time of screening, they would be excluded from the trial.
13. Any underlying medical condition that, in the Principal Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity determination or adverse events, or renders the patient ineligible to be on study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieving a CCCA defined as a reduction in the proportion of cells staining positive for Ki67 as assessed by immunohistochemistry to less than a natural logarithm, or ≤2.7%, at the post-treatment specimen. | presurgical window (period from diagnosis to surgery window of 3-6 weeks)
  Tumor's viable plus necrotic tissue, at the post-treatment specimen.

SECONDARY OUTCOMES:
The proportion of patients that achieved a complete pathologic response on surgical pathology as measured by the residual cancer burden index | presurgical window (period from diagnosis to surgery of 3-6 weeks)
  Assessed by the local pathologist at the time of definitive surgery in subjects with breast cancer
Immunohistochemical and gene expression markers of necrosis, apoptosis and tumor proliferation pathways. | presurgical window (period from diagnosis to surgery of 3-6 weeks)
  Comparison of pre (diagnostic biopsy) and post treatment (surgical resection) samples
Markers of immunomodulation including macrophages, NK, DC, CD4 T-cells, CD8 T-cells, regulatory T-cells. | presurgical window (period from diagnosis to surgery of 3-6 weeks)
  Comparison of pre (diagnostic biopsy) and post treatment (surgical resection) samples
Adverse effects of INT230-6 injected to breast cancers in healthy patients prior to surgery. | presurgical window (period from diagnosis to surgery of 3-6 weeks)
  overall safety of INT230-6 injected prior to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Angel Arnaout, MD, Principal Investigator — Ottawa Hospital Research Institute; Arif Awan, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital Research Institute and Cancer Center, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No